CLINICAL TRIAL: NCT01875978
Title: Clinical Study of Phytosterols for Insulin-like Growth Factor-1 and Endothelial Progenitor Cell Levels in Patients With Nonalcoholic Fatty Liver Disease
Brief Title: Effect of Phytosterols on Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: DMR101-IRB2-036
Record Dates: First submitted 2013-06-03; First posted 2013-06-12 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-05

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Phytosterols; Endothelial progenitor cells
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phytosterols & placebo (Active Comparator): Group A:daily 1.8g phytosterols powder for 4 weeks first;group B:placebo for 4 weeks first
  Interventions: Dietary Supplement: Phytosterols & placebo

INTERVENTIONS:
Dietary Supplement: Phytosterols & placebo — Group A:Phytosterols 1.8g/day with one meal for 4 weeks first;group B:placebo first

SUMMARY:
Phytosterols are plant sterols . Phytosterols have anti-inflammation effect. Investigators have a hypothesis: phytosterols reduce oxidative stress , enhance Insulin-like growth factor-1(IGF-1) and endothelial progenitor cells(EPCs). Therefore, phytosterols has novel role in cardiovascular protection.

DETAILED DESCRIPTION:
Fatty liver is the hepatic feature of metabolic syndrome. Metabolic syndrome increase the risk of atherosclerosis and cardiovascular disease. Adipose tissue secrete adipocytes accumulate in the liver result in fatty liver. Excess fat become low density lipoprotein-cholesterol(LDL-C) from liver. Oxidized- LDL-C adherence in the vessel result in atherosclerosis via inflammation and immune response.

Phytosterols are present in the nuts, plant oil, broccoli and so on. The structure of phytosterols are similar with cholesterols. After the competition, the smaller absorption of cholesterols. Studies showed the average consumptions of phytosterols were 200mg daily but the enough amount for cardiovascular protection of phytosterols were 2000mg daily.

Daily 2000mg phytosterols inhibit the absorption of intestine, reduce the LDL-C about 7-10%. Besides, phytosterols have the effect of anti-inflammation and anti-immune response. The anti-inflammation effect obvious inhibit the monocyte to transform to macrophage, inhibit the formation of foam cell.

Clinical studies divided into two groups: 20/20 patients and 4 weeks follow up with cross-over test.First group A: Phytosterols 1800mg/day for 4 weeks ,washout 2 weeks, then placebo 4 weeks. Another group B: placebo 4 weeks, washout 2 weeks, then phytosterols 4 weeks.Cross-over, double blind study was designed.

Investigators check the possible benefits of LDL-C, Total -cholesterol,anti-oxidant capacity,C reactive protein,insulin-like growth factor-1, endothelial progenitor cells ; the possible side effect including liver function,muscle enzyme .

ELIGIBILITY:
Inclusion Criteria:

* (1)25-80 years
* (2)Fatty liver was diagnosed by abdominal echo by the same gastrologist, review by another gastrologist

Exclusion Criteria:

* (1)Serological markers of hepatitis B virus(hepatitis B surface antigen and anti-HBs antibody) and hepatitis C virus infection (anti-HCV antibody)
* (2)Autoimmune liver disease or alcoholic liver disease(alcohol intake more than 20g per day by using a questionnaire)
* (3)Malignant diseases
* (4)Pregnancy or breast feeding
* (5)Clinical evidence of angina, congestive heart failure, valvular heart disease, inflammatory disease or thyroid dysfunction

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dalong Chen, M.D., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study from Oct. to Dec.2012 in China Medical University Hospital -Taipei branch Initially,51 patients screened .Finally, 40 patients were enrolled.
Pre-assignment Details: Statins, red yeast rice, omega-3 ,fibrates were excluded.
Groups:
- Group A:Phytosterols-placebo: phytosterols 1.8g/day first, then placebo.
- Group B:Placebo-phytosterols: Placebo first, then phytosterols 1.8g/day
Period: Study 4weeks
Arm/Group | Group A:Phytosterols-placebo | Group B:Placebo-phytosterols
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Washout 2 Weeks ,Crossover Study 4 Weeks
Arm/Group | Group A:Phytosterols-placebo | Group B:Placebo-phytosterols
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Fatty liver was diagnosed by abdominal echo, except hepatitis B,C,alcohol consumption. Totally 40 patients randomized divided to group A for phytosterols-placebo sequence and group B for placebo-phytosterols sequence.
Groups:
- Group A:Phytosterols-placebo: Daily 1.8g phytosterols powder for 4 weeks, washout 2weeks, then placebo for 4 weeks
- Group B:Placebo-phytosterols: Placebo for 4 weeks, washout 2 weeks, then daily 1.8g phytosterols powder for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Group A:Phytosterols-placebo | Group B:Placebo-phytosterols | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (12) | 51 (18) | 51 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 10 | 11 | 21
Region of Enrollment [Number; unit: participants]
  Taiwan | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Effect of Phytosterols on Patients With Nonalcoholic Fatty Liver Disease
Description: 1. Check serum metabolic status: levels in total cholesterol, low density lipoprotein-cholesterol, fasting glucose
  2. Check serum anti-inflammatory status: levels in C reactive protein
  Mid-point: end of first intervention (Group A: after phytosterols, Group B: after placebo) End-point: end of second intervention (Group A: after placebo, Group B: after phytosterols)
Time Frame: after 4 weeks phytosterols 1.8g/day
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Group A:Phytosterols-placebo | Group B:Placebo-phytosterols
Number analyzed (Participants) | 20 | 20
mg/dl
  total cholesterol (baseline) | 184.1 (6.54) | 191.65 (8.74)
  total cholesterol (mid-point) | 174.60 (6.13) | 199.25 (6.70)
  total cholesterol (end-point) | 180.55 (5.59) | 188.60 (6.03)
  low density lipoprotein (baseline) | 110.33 (6.19) | 118.45 (7.86)
  low density lipoprotein (mid-point) | 100.76 (5.96) | 121.29 (6.10)
  low density lipoprotein (end-point) | 107.54 (5.05) | 112.66 (5.46)
  fating glucose (baseline) | 106.23 (2.40) | 105.01 (1.80)
  fasting glucose (mid-point) | 100.78 (1.88) | 104.88 (2.04)
  fasting glucose (end-point) | 105.44 (2.36) | 101.65 (1.57)
  c reactive protein (baseline) | 0.32 (0.07) | 0.24 (0.05)
  c reactive protein (mid-point) | 0.23 (0.03) | 0.26 (0.04)
  C reactive protein (end-point) | 0.23 (0.03) | 0.19 (0.02)
Statistical Analysis 1: Comparison: Group A:Phytosterols-placebo vs Group B:Placebo-phytosterols; Hypothesis: phytosterols improve metabolic status; Test type: Superiority or Other; p < 0.05, t-test, 1 sided — P-value <0.05 is significance meaningful; Student's t-test, 1 sided

2. Primary Outcome: Anti-oxidative Capacity of Phytosterols on Patients With Fatty Liver Disease
Description: Check serum anti-oxidative capacity, especially the serum superoxide dismutase (SOD) levels.Serum SOD provide the anti-oxidative capacity in lipid oxidation.
  Mid-point: end of first intervention (Group A: after phytosterols, Group B: after placebo) End-point: end of second intervention (Group A: after placebo, Group B: after phytosterols)
Time Frame: after 4 weeks phytosterols 1.8g/day
Measure: Mean (Standard Error); unit: U/mg-protein
Arm/Group | Group A:Phytosterols-placebo | Group B:Placebo-phytosterols
Number analyzed (Participants) | 20 | 20
U/mg-protein
  Serum SOD (baseline) | 97.33 (2.67) | 99.41 (2.39)
  Serum SOD (mid-point) | 104.91 (3.16) | 95.1 (2.82)
  Serum SOD (end-point) | 103.28 (4.18) | 106.54 (3.76)
Statistical Analysis 1: Comparison: Group A:Phytosterols-placebo vs Group B:Placebo-phytosterols; Hypothesis: phytosterols increase the anti-oxidative capacity; Test type: Superiority or Other; p < 0.05, t-test, 1 sided — P value <0.05 for statistical significance; Student's t test, 1 sided

3. Primary Outcome: Insulin-like Growth Factor-1 Effect of Phytosterols on Patients With Nonalcoholic Fatty Liver Disease
Description: Check serum Insulin-like growth factor-1 levels. Serum Insulin-like growth factor-1 (IGF-1) influence metabolic status and reduce EPCs apoptosis via IGF-1 receptor.
  Mid-point: end of first intervention (Group A: after phytosterols, Group B: after placebo) End-point: end of second intervention (Group A: after placebo, Group B: after phytosterols)
Time Frame: after 4 weeks phytosterols 1.8g/day
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Group A:Phytosterols-placebo | Group B:Placebo-phytosterols
Number analyzed (Participants) | 20 | 20
ng/ml
  Serum IGF-1 (baseline) | 137.14 (8.36) | 153.30 (10.44)
  Serum IGF-1 (mid-point) | 167.96 (9.42) | 150.26 (9.37)
  Serum IGF-1 (end-point) | 165.23 (7.78) | 178.04 (10.88)
Statistical Analysis 1: Comparison: Group A:Phytosterols-placebo vs Group B:Placebo-phytosterols; Phytosterols increase IGF-1; Test type: Superiority or Other; p < 0.05, t-test, 1 sided — P<0.05 for statistical significance; Student's t test, 1 sided

4. Primary Outcome: Endothelial Protective Effect of Phytosterols on Patients With Non-alcoholic Fatty Liver Disease
Description: Ceck serum endothelial progenitor cells in the monocytes group but not in the lymphocytes group. Serum EPCs in the monocytes group provide the effect of endothelial repair to support novel vessel protection.
  Cytometry flow check 150,000 cells per time including monocytes and lymphocytes group. Positive cells is the EPCs in the monocytes group. Stain with KDR, call kinase insert domain receptor, also call as VEGF receptor-2.
  Mid-point: end of first intervention (Group A: after phytosterols, Group B: after placebo) End-point: end of second intervention (Group A: after placebo, Group B: after phytosterols)
Time Frame: after 4 weeks phytosterols 1.8g/day
Measure: Mean (Standard Error); unit: positive cells/150,000 cells
Arm/Group | Group A:Phytosterols-placebo | Group B:Placebo-phytosterols
Number analyzed (Participants) | 20 | 20
positive cells/150,000 cells
  EPCs with CD34+ (baseline) | 13.5 (2.38) | 18.4 (2.58)
  EPCs with CD34+ (mid-point) | 23.35 (4.88) | 18.4 (3.74)
  EPCs with CD34+ (end-point) | 18.7 (2.31) | 28.25 (3.68)
  EPCs with CD34+,KDR+ (baseline) | 0.9 (0.26) | 1.2 (0.31)
  EPCs with CD34+,KDR+ (mid-point) | 2.5 (0.34) | 1.1 (0.16)
  EPCs with CD34+,KDR+ (end-point) | 2.05 (0.23) | 2.5 (0.4)
  EPCs with KDR+,CD133+ (baseline) | 0.8 (0.24) | 1.1 (0.3)
  EPCs with KDR+,CD133+ (mid-point) | 2.45 (0.31) | 1.1 (0.16)
  EPCs with KDR+,CD133+ (end-point) | 1.9 (0.26) | 2.4 (0.42)
Statistical Analysis 1: Comparison: Group A:Phytosterols-placebo vs Group B:Placebo-phytosterols; Hypothesis:phytosterols increase endothelial progenitor cells to provide endothelial repair and vessel protection; Test type: Superiority or Other; p < 0.05, t-test, 1 sided — P value <0.05 for statistical significance; Student's t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 2 months
Description: study 4 weeks, washout 2 weeks, then cross over study 4 weeks
Groups:
- Group A: Phytosterols-placebo: Daily 1.8g phytosterols powder for 4 weeks, washout 2 weeks, then placebo for 4 weeks
- Group B: Placebo-phytosterols: placebo for 4 weeks, washout 2 weeks. then daily 1.8 g phytosterols for 4 weeks
Arm/Group | Group A: Phytosterols-placebo | Group B: Placebo-phytosterols
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Phytosterols-placebo (N=20) | Group B: Placebo-phytosterols (N=20)
Serious adverse event in the end of first intervention (Vascular disorders) | 0 (0) | 0 (0) — Group A : after phytosterols, Group B: after placebo
Serious adverse event in the end of second intervention (Vascular disorders) | 0 (0) | 0 (0) — Group A: after placebo, Group B: after phytosterols
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Phytosterols-placebo (N=20) | Group B: Placebo-phytosterols (N=20)
diarrhea in the end of first intervention (Gastrointestinal disorders) | 1 (1) | 0 (0) — Group A: after phytosterols, Group B: after placebo
diarrhea in the end of second intervention (Gastrointestinal disorders) | 0 (0) | 0 (0) — Group A: after placebo, Group B: after phytosterols

LIMITATIONS AND CAVEATS:
1. The sample size of this study is small amount
2. Abdominal ultrasound related nonalcoholic fatty liver disease diagnosis is not compatible completely

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less